CLINICAL TRIAL: NCT05032963
Title: Neurocognition After Perturbed Sleep (NAPS)
Brief Title: Neurocognition After Perturbed Sleep
Acronym: NAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Kimhy, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GCO 20-1697; 1R21MH126357 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Sleep; Cognition; Mood; Emotion Regulation; Functioning; Psychosis
MeSH Terms: conditions — Schizophrenia; Emotional Regulation; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The neurocognitive evaluators who administer the neurocognitive battery (MCCB) will be blinded to sleep schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undisturbed Sleep (Active Comparator): 8 hours sleep - Subjects randomized to the undisturbed sleep will be instructed to go to sleep at 11pm, and awoken at 7am.
  Interventions: Behavioral: Overnight polysomnography examinations
- Restricted Sleep (Experimental): 4 hours sleep - Subjects randomized to the restricted sleep will be instructed to go to sleep at 3am and awoken at 7am.
  Interventions: Behavioral: Overnight polysomnography examinations

INTERVENTIONS:
Behavioral: Overnight polysomnography examinations — sleep lab for overnight polysomnography examinations

SUMMARY:
Individuals with schizophrenia display a wide range of neurocognitive difficulties resulting in functional impairment and disability. Extensive evidence indicates insomnia and sleep disturbances play a substantial role in degrading cognitive functioning. However, the putative impact of insomnia and sleep disturbances on neurocognition and daily functioning has not been investigated in people with schizophrenia. The goal of this study is to characterize sleep in individuals with schizophrenia and quantify its impact on neurocognition and daily functioning.

DETAILED DESCRIPTION:
Individuals with SZ display a broad range of neurocognitive difficulties that have been identified as major determinants of poor functioning and disability, thus representing an important public health concern and a focal target for interventions. Extensive research literatures converge in highlighting the critical role insomnia and sleep disturbances play in degrading neurocognitive functioning. Such sleep disturbances result in clinical presentations similar to neurocognitive difficulties commonly observed in people with SZ. While insomnia and sleep disturbances are highly prevalent in people with SZ, there are scant data on the impact of sleep disturbances on neurocognition in SZ, and no data quantifying their influence on daily functioning. Thus, sleep disturbances remain poorly understood and modeled in SZ, their impact is rarely considered in clinical trials, and they remain largely unaddressed by clinicians. To address this gap in knowledge, the primary aim of this study is to characterize sleep in individuals with SZ and quantify its impact on neurocognition and daily functioning. Employing an experimental, within-person, repeated assessment design, the study team will characterize sleep architecture, duration, and quality along with cognitive, electrophysiological, biomarkers and daily functioning sequelae in 40 individuals with SZ. Participants will first complete a week-long, in-home characterization of sleep duration and quality using actigraphy and a sleep diary. Next, they will complete two overnight polysomnography examinations employing two sleep schedules:

1) undisturbed sleep; and 2) restricted sleep (4 hours). As part of these assessments, participants will provide blood samples for biomarkers analyses and complete EEG-indexed memory tasks pre- and post-sleep, along with a post-sleep battery of neurocognitive functioning.

Finally, participants will complete a 3-day ambulatory assessment using actigraphy and smartphones to explore the impact of each sleep schedule on "real-world" daily functioning including symptoms, emotion regulation, and mood.

ELIGIBILITY:
Inclusion Criteria:

* Females or males age 18-60 years
* DSM-5 diagnosis of schizophrenia, schizoaffective, or schizophreniform disorder
* Taking antipsychotic medication for >7 weeks and on current doses for 4 weeks, and/or injectable depot antipsychotics with no change in the last 3 months
* Capacity to understand all the potential risks and benefits of the study.

Exclusion Criteria:

* DSM-5 alcohol/substance diagnosis (except nicotine) within the last 6 months
* Taking medications affecting sleep propensity or architecture (other than antipsychotic medication)
* Initiation of medications known to impact cognition in previous 4 weeks or any change in doses during this period
* History of seizures/head trauma with loss of consciousness (>10 min) resulting in cognitive sequelae
* Medical or neurological conditions that could interfere with participation (e.g., untreated hypothyroidism
* Mental retardation
* Narcolepsy
* REM behavior disorder, parasomnias)
* Pregnant/ nursing
* Serious homicidal/suicidal risk (past 6 months)
* Moderate or more severe disorganization (PANSS≥4)
* Poor English reading ability (WTAR<7)
* Individuals employed as vehicle drivers/train operators or have occupations in which lapses in sustained vigilance would compromise safety
* Night shift workers or those with irregular sleep-wake rhythms (based on the week-long home actigraphy; i.e., average bedtime of 11pm±2 hours)
* Participation in the past 3 months in cognition study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery (MCCB) | Day 2, immediate upon wakening
  The composite score of the MATRICS Consensus Cognitive Battery (MCCB) will serve as a primary neurocognitive outcome. Neurocognitive functioning is indexed on the MCCB via T scores, with a mean of 50 and a SD of 10. Thus, higher scores indicate better neurocognitive performance, with T-scores of 70+ (i.e., 2 SD's over the mean) suggestive of exceptionally strong neurocognitive abilities.
MATRICS Consensus Cognitive Battery (MCCB) | Day 16, immediate upon wakening
  The composite score of the MATRICS Consensus Cognitive Battery (MCCB) will serve as a primary neurocognitive outcome. Neurocognitive functioning is indexed on the MCCB via T scores, with a mean of 50 and a SD of 10. Thus, higher scores indicate better neurocognitive performance, with T-scores of 70+ (i.e., 2 SD's over the mean) suggestive of exceptionally strong neurocognitive abilities.
Polysomnography | Days 1-2 during restricted sleep and undisturbed sleep
  Polysomnography will be used to characterize sleep including - latency, duration, continuity, and architecture assessed during over a night sleep.
Polysomnography | Days 15-16 during restricted sleep and undisturbed sleep
  Polysomnography will be used to characterize sleep including - latency, duration, continuity, and architecture assessed during over a night sleep.

CONTACTS AND LOCATIONS:
Overall Officials: David Kimhy, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Informed Consent Form (ICF) Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. The type of analysis would be to achieve aims in the approved proposal. Data will be made available by contacting the PI via email.

REFERENCES:
- [Result] Kimhy D, Ospina L, Beck-Felts K, Fakhoury A, Mullins AE, Varga AW. The Impact of Sleep on Neurocognition and Functioning in Schizophrenia-Is It Time to Wake-Up? J Psychiatr Brain Sci. 2022;7:e220001. doi: 10.20900/jpbs.20220001. Epub 2022 Jan 25. PMID 35224206